CLINICAL TRIAL: NCT03869580
Title: Incidence and Factors Associated With Double-J Urinary Stent Infection (IJJ)
Acronym: IJJ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/396
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-02

CONDITIONS: Double J Stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stent infection: Patients diagnosed with urinary tract infection associated with double J stent
- No stent infection: Patients with double J stent without infection during the study period

SUMMARY:
The aim of the study was to determine the incidence and factors associated with double-J urinary stent infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a double-J stent placement or change in the hospital

Exclusion Criteria:

* renal transplants less than one year old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a double-J stent placement or change in the hospital will be included.
  Follow-up will be repeated at 1, 3 and 6 months and urinary tract infection will be reported
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with urinary tract infection associated with double J stent | 6 months
  Number of patients with urinary tract infection associated with double J stent
Number of patients with specific clinical data associated with urinary tract infection associated with double J stent | 6 months
  Clinical data (Age, sex, gender, comorbidities, indication of procedure, duration of double J stent placement) will be compared between patient with urinary tract infection and no urinary tract infection associated with double J stent

SECONDARY OUTCOMES:
Number of patients with relapse and/or recurrence after a first urinary tract infection | 6 months
  Number of patients with relapse and/or recurrence after a first urinary tract infection

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France